CLINICAL TRIAL: NCT04756830
Title: An Open-label Uncontrolled Study to Assess the Safety and Immunogenicity of the Inactivated Adsorbed Vaccine Against COVID-19 (Coronavac) in Individuals Over 18 Years of Age During 24 Months of Follow-up
Brief Title: A Study to Assess the Safety and Immunogenicity of the Coronavac Vaccine Against COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Butantan Institute (Other Government)
Responsible Party: Principal Investigator, Jose Cerbino Neto, Senior Researcher, D'Or Institute for Research and Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IDOR_VAC_01
Record Dates: First submitted 2021-02-15; First posted 2021-02-16 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Vaccines; sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccination (Other): All participants will receive two doses of the inactivated adsorbed vaccine against COVID-19.
  Interventions: Biological: Adsorbed COVID-19 (inactivated) Vaccine

INTERVENTIONS:
Biological: Adsorbed COVID-19 (inactivated) Vaccine — Participants will receive two doses with 14-days interval of adsorbed COVID-19 (inactivated) vaccine
  Other Names: CoronaVac

SUMMARY:
This is an open-label uncontrolled study in which all participants will receive two doses of the inactivated adsorbed vaccine against COVID-19, and will be followed up for safety and immunogenicity analysis for 24 months.

DETAILED DESCRIPTION:
This is an open-label uncontrolled study in which all participants will receive two doses of the inactivated adsorbed vaccine against COVID-19, and will be followed up for safety and immunogenicity analysis for 24 months. This study will assess safety and immunogenicity of the inactivated vaccine adsorbed against COVID-19 (CoronaVac) in a population of healthy individuals older than 18 years of age.

The estimated number of participants is 1200. Participants will be recruited within 3-4 months. The total duration of the study is estimated to be 30 months after recruitment begins.

The participants will remain in the study for approximately 24 months. The study will be carried out at the clinical research center of the D'Or Institute for Research and Education (IDOR) located at the Hospital Glória D'Or, in the city of Rio de Janeiro, RJ, Brazil

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older;
* Agree with study procedures after reading and signing the Informed Consent Form

Exclusion Criteria:

* Pregnancy (confirmed by positive β-hCG test), breastfeeding and / or expressing intention to have sexual practices with reproductive potential without using contraceptive methods in the three months following vaccination
* Evidence of uncontrolled neurological, cardiac, pulmonary, hepatic or renal disease, according to anamnesis or physical examination. Significant changes in treatment or hospitalizations due to worsening of the condition in the last three months are indicators of uncontrolled disease;
* Diseases with impaired immune system including: neoplasms (except basal cell carcinoma), congenital or acquired immunodeficiencies and autoimmune diseases not controlled according to anamnesis or physical examination. Significant changes in treatment or hospitalizations due to worsening of the condition in the last three months are indicators of uncontrolled disease;
* Behavioral, cognitive or psychiatric illness that, in the opinion of the principal investigator or his medical representative, affects the participant's ability to understand and collaborate with the requirements of the study protocol
* Any alcohol or drug abuse in the last 12 months prior to inclusion in the study that has caused medical, professional or family problems, as indicated by clinical history;
* History of severe allergic reaction or anaphylaxis to the vaccine or components of the study vaccine;
* History of asplenia;
* Participation in another clinical trial with product administration under investigation during the six months prior to its inclusion in the study or scheduled participation in another clinical trial in the two years following inclusion;
* Previous participation in a COVID-19 vaccine evaluation study or previous exposure to a COVID-19 vaccine;
* Use of immunosuppressive therapies six months prior to inclusion in the study or its scheduled use within two years of inclusion. Immunosuppressive therapies will be considered: antineoplastic chemotherapy, radiation therapy, immunosuppressants to induce tolerance to transplants, among others.
* Have received an immunosuppressive dose of corticosteroids in the last three months prior to inclusion in the study or scheduled administration of an immunosuppressive dose of corticosteroids for the three months following inclusion in the study. The dose of corticosteroids considered immunosuppressive is equivalent to prednisone at a dose of 20 mg / day for adults, for more than a week. The continuous use of topical or nasal corticosteroids is not considered immunosuppressive;
* Have received blood products (transfusions or immunoglobulins) in the last three months before inclusion in the study, or scheduled administration of blood products or immunoglobulin in the two years following inclusion in the study;
* Suspected or confirmed fever within 72 hours prior to vaccination or axillary temperature greater than 37.8 ° C * on the day of vaccination (inclusion may be postponed until the participant completes 72 hours without fever);
* Possible or confirmed case of COVID-19 on the day of vaccination (vaccination can be postponed until the participant completes 72 hours without symptoms or the diagnosis is ruled out);
* Have received vaccine with live attenuated virus in the last 28 days or inactivated vaccine in the last 14 days prior to their inclusion in the study, or have immunization scheduled for the first 28 days after their inclusion in the study;
* History of bleeding disorders (for example, deficiency of clotting factors, coagulopathy, platelet dysfunction), or previous history of bleeding or significant bruising after IM injection or venipuncture.
* Any other condition that, in the opinion of the principal investigator or his medical representative, could jeopardize the safety or rights of a potential participant or that would prevent him from complying with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of local and systemic adverse reactions in the first 7 days after immunization | Seven days after each immunization
  Frequency of solicited and unsolicited local and systemic adverse reactions in the first 7 days after vaccination per age group (18-59 years old and 60 years old or older), attributed to the vaccine after causality assessment
Seroconversion rates | Two weeks after the second immunization
  Seroconversion rates in the second week after the second dose of the vaccine per age group (18-59 years and 60 years old or older).

SECONDARY OUTCOMES:
Frequency of adverse reactions up to 28 days after immunization | 28 days after the second immunization
  Frequency of unsolicited local and systemic adverse reactions up to 28 days after the second dose of the vaccine per age group (18-59 years old and 60 years old or older), attributed to the vaccine after causality assessment
Frequency of severe adverse events | Up to 12 months after first immunization
  Frequency of severe adverse events after vaccination, attributed to the vaccine after causality assessment
Frequency of adverse events of special interest | Up to 12 months after first immunization
  Frequency of adverse events of special interest after receiving, at least, one dose of the vaccine
Cell-mediated immune response | At inclusion and 4 weeks after the second vaccination
  Cell-mediated immune response at inclusion and four weeks after the second vaccination per age group (18-59 years old and 60 years old or older).
Frequency of detection of antibodies against SARS-CoV-2 | At inclusion, and two weeks, 6 months, 12 months, 18 months and 24 months after the second vaccination
  Frequency of detection of antibodies against SARS-CoV-2 at inclusion, and two weeks, 6 months, 12 months, 18 months and 24 months after the second dose of the vaccine against COVID-19.
Geometric mean titer of neutralizing antibodies | At inclusion, and two weeks, 6 months, 12 months, 18 months and 24 months after the second vaccination
  Geometric mean titer of neutralizing antibodies against SARS-CoV-2 at inclusion, and two weeks, 6 months, 12 months, 18 months and 24 months after the second dose of the vaccine against COVID-19.

OTHER OUTCOMES:
Frequency of confirmed cases of COVID-19 | Up to 24 months after inclusion
  Frequency of confirmed cases of COVID-19 per age group (18-59 years old and 60 years old or older) over 24 months.
Frequency of SARS-CoV-2 variants of concern (VOC) | Up to 24 months after inclusion
  Frequency of SARS-CoV-2 variants of concern (VOC) in confirmed cases of COVID-19.
Humoral and cellular immune response | Up to 24 months after inclusion
  Humoral and cellular immune response in confirmed cases of COVID-19

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital Gloria D'Or - Hospitais Integrados da Gavea S/A, Rio de Janeiro
  - D'Or Institute for Research and Education, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No